CLINICAL TRIAL: NCT01436773
Title: Identification of Carotid Vasa Vasorum and Correlation With Acute Coronary Events
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Flordeliza Villanueva, Professor of Medicine, University of Pittsburgh School of Medicine; Vice Chair for Pre-Clinical Research, Department of Medicine; Director, Non Invasive Cardiac Imaging; Director, Center for Ultrasound Molecular Imaging and Therapeutics, University of Pittsburgh
Other Study IDs: CVV-ACE-01
Record Dates: First submitted 2011-09-13; First posted 2011-09-20 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Recent Acute Coronary Event: Patients admitted to the hospital for recent STEMI or NSTEMI.
- Stable Coronary Artery Disease: Patients with known Coronary Artery Disease without recent acute coronary event.
- No Coronary Artery Disease: Patients with no evidence of coronary artery disease, assessed by coronary angiography.

SUMMARY:
Adventitial vasa vasorum (VV) as well as intraplaque microvessels are known to be associated with atherosclerotic plaque vulnerability. Contrast-enhanced ultrasound has been validated as a technique to measure the density of VV. Previous studies have demonstrated a relationship between identification of VV and relationship to vascular events such as stroke and myocardial infarction. No previous study has reported the utilization of contrast-enhanced ultrasound identification of VV in the carotid bed as a means of identifying patients at high risk for acute coronary events.

Aims: In this study, the investigators will aim to identify VV and intraplaque microvessels along with carotid intima media thickness (CIMT), a known marker for acute coronary events. The investigators will attempt to measure the correlation of VV with acute coronary events independent of traditional cardiovascular disease (CVD) risk factors and CIMT.

Methods: 90 volunteers (30 low risk patients, 30 patients with established coronary artery disease (CAD), and 30 patients with recent acute coronary syndrome (ACS)) will be enrolled. All patients will undergo contrast-enhanced ultrasound imaging of their carotid arteries and measurement of CIMT while obtaining baseline histories and assessment of traditional risk factors for coronary artery disease. VV density and CIMT will be measured in all patients. Statistical differences in VV among the three groups will be assessed and analyses will be made to attempt to identify if VV in the carotid bed is an independent predictor of acute coronary events after controlling for CIMT and traditional risk factors.

Study population: The study population will reflect the patient population of UPMC. No individual will be excluded on the basis of race, gender, or ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred for elective left heart catheterization in the past three months or individuals who have undergone recent left heart catheterization for acute coronary syndrome in the past 3 months

Exclusion Criteria:

* Inability to provided informed consent
* Pregnancy or of lack confirmed urine or serum B-hcg testing in pre-menopausal women under the age of 50
* Known allergy to Definity (registered trademark)
* Contraindications to Definity including permanent or transient right to left or bidirectional cardiac shunts, allergy to perflutren, severe pulmonary hypertension
* Known cocaine abuse within the past year
* History of heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented coronary artery disease and/or recent acute coronary event who undergo left heart catheterization, and patients with history and previous testing that cannot rule out coronary artery disease and undergo elective left heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Carotid Artery Adventitial Vaso Vasorum Density | Measured within 1 week of enrollment.
  Assessed with ultrasound contrast agent, Definity, from Lantheus Medical Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Flordeliza Villanueva, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States